CLINICAL TRIAL: NCT02277015
Title: Pediatric Tracheal Intubation Using Four Video-laryngoscopes and the Miller Laryngoscope With and Without Chest Compressions
Brief Title: Intubation During Pediatric Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ETI/2014/02
Record Dates: First submitted 2014-10-26; First posted 2014-10-28 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-10

CONDITIONS: Cardiac Arrest; Endotracheal Intubation; Pediatric Manikin
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI without chest compressions (Experimental): Endotracheal intubation during pediatric resuscitation without chest compressions.
  Interventions: Device: Miller Laryngoscope; Device: The Berci-Kaplan DCI; Device: The AirTraq; Device: GlideScope GVL; Device: The Pentax AWS
- ETI with chest compressions (Experimental): Endotracheal intubation during pediatric resuscitation with chest compressions. Chest compression was performed using LUCAS-2 (Physio-Control).
  Interventions: Device: Miller Laryngoscope; Device: The Berci-Kaplan DCI; Device: The AirTraq; Device: GlideScope GVL; Device: The Pentax AWS

INTERVENTIONS:
Device: Miller Laryngoscope — Direct Laryngoscopy
Device: The Berci-Kaplan DCI — Videolaryngoscope-1
Device: The AirTraq — Videolaryngoscope-2
Device: GlideScope GVL — Videolaryngoscope-3
Device: The Pentax AWS — Videolaryngoscope-4

SUMMARY:
The European Resuscitation Council (ERC) 2010 cardiopulmonary resuscitation (CPR) guidelines suggest that intubators should be able to secure the airway without interrupting chest compression. We examine the performance of the Berci-Kaplan DCI (BERCI), the GlideScope (GVL), the AirTraq, the Pentax AWS (Pentax) and the Miller laryngoscope (MIL) for endotracheal intubation (ETI) during pediatric resuscitation with and without chest compressions.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medicine personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Intubation Time | 1 month
  time in seconds required for a successful intubation attempt with the five different ETI devices

SECONDARY OUTCOMES:
Successful intubation | 1 month
  effectiveness of first, second, third intubation attempts and overall effectiveness intubation attempt using all intubation devices
POGO score | 1 month
  self reported percentage og glottis opening (POGO) score
VAS score | 1 month
  To assess subjective opinion about the difficulty of the procedure, participants were asked to rate it on a visual analogue scale (VAS) with a score from 1 (very easy) to 5 (very difficult).
Preferred ETI device | 1 month
  participants were asked which method of ETI they would prefer in a real-life resuscitation.
First Pass Attempt | 1 month
  Endotracheal Intubation (ETI) attempt will be defined as tip of the laryngoscope blade passing the patient's lips. First attempt success rate will be defined as the number of successful placements occurring on the first attempt to place the endotracheal tube.
Overall Success | intraoperative
  Overall success rate will be defined as the total number of successful placements divided by the total number of patients treated.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland